CLINICAL TRIAL: NCT01775878
Title: A Randomized Study Comparing Usual Diabetes Care Management to Telemetric Home-based Monitoring of Glucose and Blood Pressure in Patients With Diabetes (TELEGAP)
Brief Title: Diabetes Care Management Trial of Telemetric Monitoring
Acronym: TELEGAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CN-08JMink-01
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes
Keywords: Diabetes; HbA1c; Fructosamine; Blood Pressure; Telemonitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): This arm received usual care from the diabetes care managers
- Telemonitoring Device (Experimental): Patients in this arm received a telemonitoring device installed in their homes
  Interventions: Device: Telemonitoring Device

INTERVENTIONS:
Device: Telemonitoring Device — Telemonitoring device was installed in patients' homes
  Other Names: Samsung Health Diary
  Arms: Telemonitoring Device

SUMMARY:
The study is a two-arm, parallel-comparison, single-blind, randomized controlled trial, and will be offered to Kaiser Permanente members aged 18 - 75 years old who present to the Santa Rosa Diabetes Care Management Center with Type 2 diabetes mellitus. Participants will be randomly assigned to one of two treatment arms. The telemedicine group or the group receiving usual care (the control group).

This study hopes to show the usefulness of this telemonitoring technology and more specifically, to assess whether this device improves markers of control of diabetes, glycemic control, and cardiovascular risk factors

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years old,
* diagnosis of type 2 diabetes mellitus for at least 1 month,
* eligible for and referred to the diabetes care management program,
* HbA1c values in the range: 7.5% to 10.5%.

Exclusion Criteria:

* Weight > 330 lbs,
* estimated glomerular filtration rate (GFR) < 45,
* unstable coronary artery disease,
* severe peripheral vascular disease which restricted exercise,
* end-stage liver disease,
* undergoing treatment for cancer,
* pregnant or not using appropriate birth control,
* no broadband internet access in their homes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Fructosamine | 6 weeks
  Change from baseline to 6 weeks in serum fructosamine levels
glycosylated hemoglobin | 6 months
  change from baseline to 6 months in serum HbA1c levels

SECONDARY OUTCOMES:
blood pressure | 6 weeks and 6 months
  goal of systolic < 130 mmHg and diastolic < 70 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Minkoff, MD, Principal Investigator — Kaiser Permanente